CLINICAL TRIAL: NCT06326554
Title: Single Arm Pilot Trial of Virtual and In-person Symptom Screening With Targeted Early Palliative Care (STEP2)
Brief Title: Pilot Trial of Virtual and In-person STEP2
Acronym: STEP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Camilla Zimmermann, Principal Investigator, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-5933
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STEP2 (Experimental): Moderate-to-severe symptoms on the Edmonton Symptom Assessment System-revised (ESAS-r+) tool will trigger an email to the study team and the study triage nurse. The study triage nurse will review the scores via electronic medical record and call the patient within 2 business days to offer immediate advice by phone. During the phone call, the study triage nurse will offer to schedule a formal in-person or virtual palliative care clinic (PCC) visit. Participants agreeing to the PCC referral subsequently receive at least monthly in-person and/or virtual PCC follow-up visits until study end, based on patient needs and care provider preference.
  Interventions: Behavioral: Virtual and in-person Symptom screening with Targeted Early Palliative care (STEP2)

INTERVENTIONS:
Behavioral: Virtual and in-person Symptom screening with Targeted Early Palliative care (STEP2) — Study nurse will offer a palliative care clinic visit referral alongside usual cancer care to participants who report moderate to high symptom burden.

SUMMARY:
The goal of this clinical trial is to assess the feasibility of offering oncology patients a referral to the outpatient palliative care clinic based on virtual symptom screening before oncology clinic appointments, and to qualitatively explore factors patients consider when deciding to accept or defer a visit to this clinic.

Participants will be asked to complete questionnaires assessing quality of life, symptom burden, depression, anxiety, and satisfaction with care at baseline, 2, 4, and 6 months.

DETAILED DESCRIPTION:
To improve equitable access to early palliative care based on symptom severity, the investigators developed Symptom screening with Targeted Early Palliative care (STEP) and demonstrated its feasibility in a previous trial. STEP was designed and tested before the COVID-19 pandemic and was based on symptom screening using tablets/computers in oncology clinics and in-person visits in the palliative care clinic. In response to changes in hospital care as a result of the COVID-19 pandemic, the investigators developed a novel, mixed in-person and virtually delivered intervention, STEP2.

The investigators propose to test STEP2 in a single-arm pilot trial, enrolling outpatients with advanced cancer and a prognosis of 6 months to 3 years. Participants will complete the Edmonton Symptom Assessment System-revised (ESAS-r+) tool electronically before oncology appointments (as is usual care in Ontario, Canada); in addition, if patients report moderate to high symptom scores, they will receive nurse-led triage and targeted referral to specialized palliative care. Quality of life, symptom burden, depression, anxiety and satisfaction with care will be assessed at baseline, 2, 4, and 6 months using questionnaires.

The objectives of this study are 1) to assess the feasibility of the STEP2 intervention, including completion of virtual symptom screening before oncology clinic appointments and completing triggered palliative care visits by video as well as in person; and 2) to explore factors patients consider when deciding to accept or defer a visit to the outpatient palliative care clinic.

ELIGIBILITY:
Inclusion Criteria:

* age 18+ years
* stage IV cancer (stage III or IV for lung or pancreas cancers; hormone-refractory for prostate and ER-positive breast cancers)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* oncologist-estimated prognosis of 6-36 months
* willingness to complete routine online symptom screening at the Princess Margaret Cancer Centre

Exclusion Criteria:

* insufficient English literacy to complete study procedures
* oncologist-determined poor cognitive status
* already received or currently receiving specialized palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2025-12-11 (Actual)

PRIMARY OUTCOMES:
FACIT-PAL 14 | 6 months
  A 14-item version of the Functional Assessment of Chronic Illness Therapy (FACIT) scale, with items that are considered relevant for patients with advanced cancer. Scoring ranges from 0-56 with lower scores indicating better quality of life.

SECONDARY OUTCOMES:
FACIT-PAL 14 | 2 and 4 months
  A 14-item version of the Functional Assessment of Chronic Illness Therapy (FACIT) scale, with items that are considered relevant for patients with advanced cancer. Scores range from 0-4 per item with higher scores indicating worse quality of life.
ESAS-r-CS | 2, 4, and 6 months
  Edmonton Symptom Assessment System-revised (ESAS-r-CS) measure with eleven scales with anchors of 0 (best) and 10 (worst) for pain, fatigue, drowsiness, nausea, anxiety, depression, appetite, dyspnea, well-being, constipation and sleep.
PHQ-9 | 2, 4, and 6 months
  A 9-item Patient Health Questionnaire (PHQ-9) for screening, diagnosing and monitoring the severity of depression. Scores range from 0-3 per item with higher scores indicating worse depression.
FAMCARE-P16 | 2, 4, and 6 months
  Modified family caregiver (FAMCARE) scale measuring patient satisfaction with information-giving, availability of care, psychological care and physical patient care in patients with advanced cancer. Scores range from 1-5 per item with higher scores indicating greater satisfaction.
Generalized Anxiety Disorder-7 | 2, 4, and 6 months
  A valid and brief 7-item Generalized Anxiety Disorder (GAD-7) tool measuring severity of anxiety in patients. Scores range from 0-3 per item with higher scores indicating worse anxiety.
Patient Global Impression of Change | 2, 4, and 6 months
  A single-item patient-reported measure assessing change in health status and efficacy of an intervention, and is a widely used clinically relevant tool across many health conditions. The scale ranges from 1-7 and higher scores indicate worse change in health status.

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Zimmermann, MD PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No